CLINICAL TRIAL: NCT04441138
Title: Phase II Trial of Concurrent, Split Course Chemoradiation Followed by Durvalumab (MEDI4736) in Poor Risk and/or Elderly Patients With Newly Diagnosed Stage III Non-small Cell Lung Cancer
Brief Title: Chemoradiation Followed by Durvalumab in Poor Risk and/or Elderly Patients With Stage III NSCLC
Acronym: ESR1814205
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Institutional constraints due to research staffing and diminished data safety monitoring infrastructure
Sponsor: Rush University Medical Center (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Gaurav Marwaha, Principal Investigator, Rush University Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR 18-14205 | 19010808
Record Dates: First submitted 2020-04-21; First posted 2020-06-22 (Actual); Results first posted 2025-05-28 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Stage III Non-small-cell Lung Cancer
Keywords: Stage III NSCLC; Durvalumab; Elderly; Poor-risk; chemoradiation
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Concurrent, Split Course Chemoradiation Followed by Durvalumab (Experimental): Concurrent, Split Course Chemoradiation Followed by Durvalumab (MEDI4736) in Poor Risk and/or Elderly Patients With Newly Diagnosed Stage III Non-small Cell Lung Cancer
  Interventions: Drug: Durvalumab

INTERVENTIONS:
Drug: Durvalumab — Adjuvant Durvalumab in Poor Risk and/or Elderly Patients With Newly Diagnosed Stage III Non-small Cell Lung Cancer who have completed concurrent, split course chemoradiation without progression of disease
  Other Names: MEDI4736; imfinzi

SUMMARY:
Elderly (age 70 years or older) or >18 years old AND poor risk (ECOG 2) newly diagnosed stage IIIA-C (AJCC 8th edition) inoperable non-small cell lung cancer (NSCLC) patients are eligible to participate in this phase II open label study of concurrent, split course chemoradiation followed by Durvalumab (MEDI4736).

DETAILED DESCRIPTION:
The rationale for the study is to identify another cohort of stage III NSCLC for whom adjuvant Durvalumab can be safely given, expanding its utilization and benefits. With a unique, extremely well-tolerated 4-phase split course CRT regimen preceding the administration of Durvalumab, we expect to be able to offer adjuvant Durvalumab to a significant proportion of patients on study.

Patients who have completed four cycles of chemoradiation (Radiation is 60 Gy in 30 fractions administered over 12 weeks with 1-1.5 week breaks between cycles; Chemotherapy is once every 3 weeks for up to 4 cycles) will go on to receive durvalumab (MEDI4736) monotherapy as 1500mg durvalumab (MEDI4736) via IV infusion Q4W for up to a maximum of 12 months (up to 13 doses/cycles) with the last administration on week 48 until confirmed disease progression unless there is unacceptable toxicity, withdrawal of consent, or another discontinuation criterion is met.

Primary objectives are:

1. To determine the percentage of poor risk and/or elderly unresectable stage III NSCLC patients who complete split course chemoradiation
2. To determine the safety and tolerability of durvalumab (MEDI4736) after completion of chemoradiation in this group of patients.

Secondary Objectives are:

1. To determine the 1-year overall survival rate
2. To determine the 1-year progression-free survival rate
3. To determine the 1-year loco-regional progression-free survival rate
4. To determine rate of grade 3 and 4 toxicities with this regimen in the selected patient population

ELIGIBILITY:
Inclusion Criteria:

1. Participants must have histologically or cytologically confirmed stage IIIA-C (AJCC 8th edition) non-small cell lung cancer, that will be treated with curative intent.
2. Participants must have been deemed medically inoperable by multidisciplinary team/tumor board
3. Participants must have been staged with a PET/CT within 30 days of enrollment
4. Patients must have undergone an MRI Brain w/IV contrast, or CT brain if MRI not feasible, confirming no evidence of brain metastases, within 30 days of enrollment.
5. Participants must be elderly (age 70 years or older and PS 0-1) or >18 years old AND poor risk (ECOG 2)
6. Participants ideally have endobronchial ultrasound biopsy (EBUS) or mediastinoscopy to confirm nodal status, but can be deferred if PET/CT imaging characteristics are highly suggestive of nodal metastases
7. Participants should have a life expectancy of >6 months
8. Participants must have normal organ and marrow function: Leukocytes >3000/mcL; ANC >1500/mcL; PLT>100000/mcL; Hemoglobin ≥9.0 g/dL
9. Serum bilirubin ≤1.5 x institutional upper limit of normal (ULN)
10. AST/ALT <2.5 x institutional upper limit of normal
11. Measured creatinine clearance (CL) >40 mL/min or Calculated creatinine CL>40 mL/min by the Cockcroft-Gault formula

    Males:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) 72 x serum creatinine (mg/dL)

    Females:

    Creatinine CL (mL/min) = Weight (kg) x (140 - Age) x 0.85 72 x serum creatinine (mg/dL)
12. Patients must be capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (eg, Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations. If study includes Japan add (For patients aged <20 years and enrolling in Japan, a written informed consent should be obtained from the patient and his or her legally acceptable representative.)
13. Body weight >30kg
14. Evidence of post-menopausal status or negative urinary or serum pregnancy test for female pre-menopausal patients. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:

    Women <50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of exogenous hormonal treatments and if they have luteinizing hormone and follicle-stimulating hormone levels in the post-menopausal range for the institution or underwent surgical sterilization (bilateral oophorectomy or hysterectomy).

    Women ≥50 years of age would be considered post-menopausal if they have been amenorrheic for 12 months or more following cessation of all exogenous hormonal treatments, had radiation-induced menopause with last menses >1 year ago, had chemotherapy-induced menopause with last menses >1 year ago, or underwent surgical sterilization (bilateral oophorectomy, bilateral salpingectomy or hysterectomy).
15. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. History of allergic reactions attributed to compounds of similar chemical or biologic composition to carboplatin, pemetrexed (for patients with adenocarcinoma), etoposide (for patients with squamous cell carcinoma), or immunotherapy
2. Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic CHF, unstable angina pectoris, cardiac arrhythmia, or psychiatric/social situations that would limit compliance with study requirements.
3. Pregnant women
4. HIV positive patients
5. Participation in another clinical study with an investigational product during the last 6 months
6. Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
7. Receipt of the last dose of anticancer therapy (CRT) ≤7 days prior to the first dose of study drug. If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca/MedImmune and the investigator
8. Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria

   1. Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
   2. Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
9. Any concurrent chemotherapy, IP, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
10. Major surgical procedure (as defined by the Investigator) within 28 days prior to the first dose of IP. Note: Local surgery of isolated lesions for palliative intent is acceptable.
11. History of allogenic organ transplantation.
12. Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). The following are exceptions to this criterion:

    1. Patients with vitiligo or alopecia
    2. Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
    3. Any chronic skin condition that does not require systemic therapy
    4. Patients without active disease in the last 5 years may be included but only after consultation with the study physician
    5. Patients with celiac disease controlled by diet alone
13. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent
14. History of another primary malignancy except for

    1. Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of IP and of low potential risk for recurrence
    2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
    3. Adequately treated carcinoma in situ without evidence of disease
15. History of leptomeningeal carcinomatosis
16. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated from 3 ECGs (within 15 minutes at 5 minutes apart) <<for durvalumab monotherapy.
17. History of active primary immunodeficiency
18. Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C, or human immunodeficiency virus (positive HIV 1/2 antibodies). Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
19. Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab. The following are exceptions to this criterion:

    1. Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
    2. Systemic corticosteroids at physiologic doses not to exceed <<10 mg/day>> of prednisone or its equivalent
    3. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
20. Receipt of live attenuated vaccine within 30 days prior to the first dose of IP. Note: Patients, if enrolled, should not receive live vaccine whilst receiving IP and up to 30 days after the last dose of IP.
21. Female patients who are pregnant or breastfeeding or male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy.
22. Known allergy or hypersensitivity to any of the study drugs or any of the study drug excipients.
23. Prior randomisation or treatment in a previous durvalumab clinical study regardless of treatment arm assignment.
24. Patients who have received prior anti-PD-1, anti PD-L1, including durvalumab or anti CTLA-4:

    1. Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
    2. All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study.
    3. Must not have experienced a ≥Grade 3 immune related AE or an immune related neurologic or ocular AE of any grade while receiving prior immunotherapy. NOTE: Patients with endocrine AE of ≤Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic.
    4. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
25. Judgment by the investigator that the patient is unsuitable to participate in the study and the patient is unlikely to comply with study procedures, restrictions and requirements.

Procedures for withdrawal of incorrectly enrolled patients are presented in Section 4.3 Withdrawal of patients from study treatment and/or study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-02-25 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaurav Marwaha, MD, Principal Investigator — Rush University Cancer Center
Locations (1):
- Rush University Cancer Center, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Kurata T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Faivre-Finn C, Reck M, Vansteenkiste J, Spigel DR, Wadsworth C, Melillo G, Taboada M, Dennis PA, Ozguroglu M; PACIFIC Investigators. Overall Survival with Durvalumab after Chemoradiotherapy in Stage III NSCLC. N Engl J Med. 2018 Dec 13;379(24):2342-2350. doi: 10.1056/NEJMoa1809697. Epub 2018 Sep 25. PMID 30280658
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Bonomi P, Blumenthal G, Ferris AS, Stewart DJ, Selig WKD, Krug LM, Allen J, Ison G, Langer CJ, Melemed A, Odogwu L, Basu Roy U, Sandler A. Making Lung Cancer Clinical Trials More Inclusive: Recommendations for Expanding Eligibility Criteria. J Thorac Oncol. 2018 Jun;13(6):748-751. doi: 10.1016/j.jtho.2018.02.013. No abstract available. PMID 29793646
- [Background] Jalal SI, Riggs HD, Melnyk A, Richards D, Agarwala A, Neubauer M, Ansari R, Govindan R, Bruetman D, Fisher W, Breen T, Johnson CS, Yu M, Einhorn L, Hanna N. Updated survival and outcomes for older adults with inoperable stage III non-small-cell lung cancer treated with cisplatin, etoposide, and concurrent chest radiation with or without consolidation docetaxel: analysis of a phase III trial from the Hoosier Oncology Group (HOG) and US Oncology. Ann Oncol. 2012 Jul;23(7):1730-8. doi: 10.1093/annonc/mdr565. Epub 2011 Dec 9. PMID 22156624
- [Background] Stinchcombe TE, Zhang Y, Vokes EE, Schiller JH, Bradley JD, Kelly K, Curran WJ Jr, Schild SE, Movsas B, Clamon G, Govindan R, Blumenschein GR, Socinski MA, Ready NE, Akerley WL, Cohen HJ, Pang HH, Wang X. Pooled Analysis of Individual Patient Data on Concurrent Chemoradiotherapy for Stage III Non-Small-Cell Lung Cancer in Elderly Patients Compared With Younger Patients Who Participated in US National Cancer Institute Cooperative Group Studies. J Clin Oncol. 2017 Sep 1;35(25):2885-2892. doi: 10.1200/JCO.2016.71.4758. Epub 2017 May 11. PMID 28493811
- [Background] Garg S, Gielda BT, Kiel K, Turian JV, Fidler MJ, Batus M, Bonomi P, Sher DJ. Patterns of locoregional failure in stage III non-small cell lung cancer treated with definitive chemoradiation therapy. Pract Radiat Oncol. 2014 Sep-Oct;4(5):342-348. doi: 10.1016/j.prro.2013.12.002. Epub 2014 Jan 16. PMID 25194104
- [Background] Gielda BT, Marsh JC, Zusag TW, Faber LP, Liptay M, Basu S, Warren WH, Fidler MJ, Batus M, Abrams RA, Bonomi P. Split-course chemoradiotherapy for locally advanced non-small cell lung cancer: a single-institution experience of 144 patients. J Thorac Oncol. 2011 Jun;6(6):1079-86. doi: 10.1097/JTO.0b013e3182199a7c. PMID 21532501
- [Background] Koshy M, Malik R, Spiotto M, Mahmood U, Rusthoven CG, Sher DJ. Association between intensity modulated radiotherapy and survival in patients with stage III non-small cell lung cancer treated with chemoradiotherapy. Lung Cancer. 2017 Jun;108:222-227. doi: 10.1016/j.lungcan.2017.04.006. Epub 2017 Apr 17. PMID 28625640
- [Background] Chun SG, Hu C, Choy H, Komaki RU, Timmerman RD, Schild SE, Bogart JA, Dobelbower MC, Bosch W, Galvin JM, Kavadi VS, Narayan S, Iyengar P, Robinson CG, Wynn RB, Raben A, Augspurger ME, MacRae RM, Paulus R, Bradley JD. Impact of Intensity-Modulated Radiation Therapy Technique for Locally Advanced Non-Small-Cell Lung Cancer: A Secondary Analysis of the NRG Oncology RTOG 0617 Randomized Clinical Trial. J Clin Oncol. 2017 Jan;35(1):56-62. doi: 10.1200/JCO.2016.69.1378. Epub 2016 Oct 31. PMID 28034064
- [Background] Alexandrov LB, Nik-Zainal S, Wedge DC, Aparicio SA, Behjati S, Biankin AV, Bignell GR, Bolli N, Borg A, Borresen-Dale AL, Boyault S, Burkhardt B, Butler AP, Caldas C, Davies HR, Desmedt C, Eils R, Eyfjord JE, Foekens JA, Greaves M, Hosoda F, Hutter B, Ilicic T, Imbeaud S, Imielinski M, Jager N, Jones DT, Jones D, Knappskog S, Kool M, Lakhani SR, Lopez-Otin C, Martin S, Munshi NC, Nakamura H, Northcott PA, Pajic M, Papaemmanuil E, Paradiso A, Pearson JV, Puente XS, Raine K, Ramakrishna M, Richardson AL, Richter J, Rosenstiel P, Schlesner M, Schumacher TN, Span PN, Teague JW, Totoki Y, Tutt AN, Valdes-Mas R, van Buuren MM, van 't Veer L, Vincent-Salomon A, Waddell N, Yates LR; Australian Pancreatic Cancer Genome Initiative; ICGC Breast Cancer Consortium; ICGC MMML-Seq Consortium; ICGC PedBrain; Zucman-Rossi J, Futreal PA, McDermott U, Lichter P, Meyerson M, Grimmond SM, Siebert R, Campo E, Shibata T, Pfister SM, Campbell PJ, Stratton MR. Signatures of mutational processes in human cancer. Nature. 2013 Aug 22;500(7463):415-21. doi: 10.1038/nature12477. Epub 2013 Aug 14. PMID 23945592
- [Background] Brahmer JR, Tykodi SS, Chow LQ, Hwu WJ, Topalian SL, Hwu P, Drake CG, Camacho LH, Kauh J, Odunsi K, Pitot HC, Hamid O, Bhatia S, Martins R, Eaton K, Chen S, Salay TM, Alaparthy S, Grosso JF, Korman AJ, Parker SM, Agrawal S, Goldberg SM, Pardoll DM, Gupta A, Wigginton JM. Safety and activity of anti-PD-L1 antibody in patients with advanced cancer. N Engl J Med. 2012 Jun 28;366(26):2455-65. doi: 10.1056/NEJMoa1200694. Epub 2012 Jun 2. PMID 22658128
- [Background] Butte MJ, Keir ME, Phamduy TB, Sharpe AH, Freeman GJ. Programmed death-1 ligand 1 interacts specifically with the B7-1 costimulatory molecule to inhibit T cell responses. Immunity. 2007 Jul;27(1):111-22. doi: 10.1016/j.immuni.2007.05.016. Epub 2007 Jul 12. PMID 17629517
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Ellis S, Carroll KJ, Pemberton K. Analysis of duration of response in oncology trials. Contemp Clin Trials. 2008 Jul;29(4):456-65. doi: 10.1016/j.cct.2007.10.008. Epub 2007 Nov 12. PMID 18187370
- [Background] Fife BT, Bluestone JA. Control of peripheral T-cell tolerance and autoimmunity via the CTLA-4 and PD-1 pathways. Immunol Rev. 2008 Aug;224:166-82. doi: 10.1111/j.1600-065X.2008.00662.x. PMID 18759926
- [Background] Hirano F, Kaneko K, Tamura H, Dong H, Wang S, Ichikawa M, Rietz C, Flies DB, Lau JS, Zhu G, Tamada K, Chen L. Blockade of B7-H1 and PD-1 by monoclonal antibodies potentiates cancer therapeutic immunity. Cancer Res. 2005 Feb 1;65(3):1089-96. PMID 15705911
- [Background] Iwai Y, Ishida M, Tanaka Y, Okazaki T, Honjo T, Minato N. Involvement of PD-L1 on tumor cells in the escape from host immune system and tumor immunotherapy by PD-L1 blockade. Proc Natl Acad Sci U S A. 2002 Sep 17;99(19):12293-7. doi: 10.1073/pnas.192461099. Epub 2002 Sep 6. PMID 12218188
- [Background] Keir ME, Butte MJ, Freeman GJ, Sharpe AH. PD-1 and its ligands in tolerance and immunity. Annu Rev Immunol. 2008;26:677-704. doi: 10.1146/annurev.immunol.26.021607.090331. PMID 18173375
- [Background] Lan and DeMets 1983 Lan KKG, DeMets DL. Discrete sequential boundaries for clinical trials. Biometrika 1983;70:659 63
- [Background] Brahmer et al. 2014 Brahmer JR, Horn L, Gandhi L, Spigel DR, Antonia SJ, Rizvi NA, et al. Nivolumab (anti PD 1, BMS-936558, ONO-4538) in patients (pts) with advanced non-small-cell lung cancer (NSCLC): Survival and clinical activity by subgroup analysis [ASCO abstract 8112]. J Clin Oncol 2014;32(Suppl).
- [Background] o Drake et al. 2013 Drake CG, McDermott DF, Sznol M, Choueiri TK, Kluger HM, Powderly JD et al. Survival, safety, and response duration results of nivolumab (Anti-PD-1; BMS-936558; ONO-4538) in a phase I trial in patients with previously treated metastatic renal cell carcinoma (mRCC): Long-term patient follow-up [abstract 4514]. J Clin Oncol 2013;31(Suppl).
- [Background] Fairman et al. 2014 Fairman D, Narwal R, Liang M, Robbins PB, Schneider A, Chavez C, et al. Pharmacokinetics of durvalumab, a fully human anti-PDL1 monoclonal antibody, in patients with advanced solid tumours. Journal of Clinical Oncology, 2014 ASCO Annual Meeting Abstracts;32(5s): (suppl; abstr 2602).
- [Background] Herbst et al. 2013 Herbst RS, Gordon MS, Fine GD, Sosman JA, Soria JC, Hamid O, et al. A study of MPDL3280A, an engineered PD-L1 antibody in patients with locally advanced or metastatic tumours [abstract 3000]. J Clin Oncol 2013;31(Suppl 15).
- [Background] Hodi et al. 2014 Hodi FS, Sznol M, Kluger HM, McDermott DF, Carvajal RD, Lawrence DP et al. Long-term survival of ipilimumab-naive patients (pts) with advanced melanoma (MEL) treated with nivolumab (anti-PD-1, BMS-936558, ONO-4538) in a Phase I trial [ASCO abstract 9002]. J Clin Oncol 2014; 32(Suppl).
- [Background] Narwal R, Roskos LK, Robbie GJ. Population pharmacokinetics of sifalimumab, an investigational anti-interferon-alpha monoclonal antibody, in systemic lupus erythematosus. Clin Pharmacokinet. 2013 Nov;52(11):1017-27. doi: 10.1007/s40262-013-0085-2. PMID 23754736
- [Background] Ng CM, Lum BL, Gimenez V, Kelsey S, Allison D. Rationale for fixed dosing of pertuzumab in cancer patients based on population pharmacokinetic analysis. Pharm Res. 2006 Jun;23(6):1275-84. doi: 10.1007/s11095-006-0205-x. Epub 2006 May 26. PMID 16715358
- [Background] Okudaira K, Hokari R, Tsuzuki Y, Okada Y, Komoto S, Watanabe C, Kurihara C, Kawaguchi A, Nagao S, Azuma M, Yagita H, Miura S. Blockade of B7-H1 or B7-DC induces an anti-tumor effect in a mouse pancreatic cancer model. Int J Oncol. 2009 Oct;35(4):741-9. doi: 10.3892/ijo_00000387. PMID 19724910
- [Background] Pardoll DM. The blockade of immune checkpoints in cancer immunotherapy. Nat Rev Cancer. 2012 Mar 22;12(4):252-64. doi: 10.1038/nrc3239. PMID 22437870
- [Background] Paterson AM, Brown KE, Keir ME, Vanguri VK, Riella LV, Chandraker A, Sayegh MH, Blazar BR, Freeman GJ, Sharpe AH. The programmed death-1 ligand 1:B7-1 pathway restrains diabetogenic effector T cells in vivo. J Immunol. 2011 Aug 1;187(3):1097-105. doi: 10.4049/jimmunol.1003496. Epub 2011 Jun 22. PMID 21697456
- [Background] Powles T, Eder JP, Fine GD, Braiteh FS, Loriot Y, Cruz C, Bellmunt J, Burris HA, Petrylak DP, Teng SL, Shen X, Boyd Z, Hegde PS, Chen DS, Vogelzang NJ. MPDL3280A (anti-PD-L1) treatment leads to clinical activity in metastatic bladder cancer. Nature. 2014 Nov 27;515(7528):558-62. doi: 10.1038/nature13904. PMID 25428503
- [Background] Qin A, Coffey DG, Warren EH, Ramnath N. Mechanisms of immune evasion and current status of checkpoint inhibitors in non-small cell lung cancer. Cancer Med. 2016 Sep;5(9):2567-78. doi: 10.1002/cam4.819. Epub 2016 Jul 15. PMID 27416962
- [Background] Rizvi et al. 2015 Rizvi N, Brahmer J, Ou S-H, Segal NH, Khleif SN, Hwu WJ. Safety and clinical activity of MEDI4736, an anti-programmed cell death-ligand-1 (PD-L1) antibody, in patients with nonsmall cell lung cancer (NSCLC). J Clin Oncol 2015;33:Abstract 8032.
- [Background] Schadendorf et al. 2013 Schadendorf D, Hodi FS, Robert C et al. Pooled analysis of long-term survival data from phase II and phase III trials of ipilimumab in metastatic or locally advanced, unresectable melanoma [abstract 24]. Presented at European Cancer Congress 2013 (ECCO-ESMO-ESTRO); 27 September to 01 October 2013; Amsterdam, The Netherlands.
- [Background] Segal et al. 2015 Segal NH, Ou S-HI, Balmanoukian AS, Fury MG, Massarelli E, Brahmer JR, et al. Safety and efficacy of MEDI4736, an anti-PD-L1 antibody, in patients from a squamous cell carcinoma of the head and neck (SCCHN) expansion cohort. J Clin Oncol 2015;33:Abstract 3011.
- [Background] Stewart R, Morrow M, Hammond SA, Mulgrew K, Marcus D, Poon E, Watkins A, Mullins S, Chodorge M, Andrews J, Bannister D, Dick E, Crawford N, Parmentier J, Alimzhanov M, Babcook JS, Foltz IN, Buchanan A, Bedian V, Wilkinson RW, McCourt M. Identification and Characterization of MEDI4736, an Antagonistic Anti-PD-L1 Monoclonal Antibody. Cancer Immunol Res. 2015 Sep;3(9):1052-62. doi: 10.1158/2326-6066.CIR-14-0191. Epub 2015 May 5. PMID 25943534
- [Background] Topalian SL, Hodi FS, Brahmer JR, Gettinger SN, Smith DC, McDermott DF, Powderly JD, Carvajal RD, Sosman JA, Atkins MB, Leming PD, Spigel DR, Antonia SJ, Horn L, Drake CG, Pardoll DM, Chen L, Sharfman WH, Anders RA, Taube JM, McMiller TL, Xu H, Korman AJ, Jure-Kunkel M, Agrawal S, McDonald D, Kollia GD, Gupta A, Wigginton JM, Sznol M. Safety, activity, and immune correlates of anti-PD-1 antibody in cancer. N Engl J Med. 2012 Jun 28;366(26):2443-54. doi: 10.1056/NEJMoa1200690. Epub 2012 Jun 2. PMID 22658127
- [Background] Topalian SL, Sznol M, McDermott DF, Kluger HM, Carvajal RD, Sharfman WH, Brahmer JR, Lawrence DP, Atkins MB, Powderly JD, Leming PD, Lipson EJ, Puzanov I, Smith DC, Taube JM, Wigginton JM, Kollia GD, Gupta A, Pardoll DM, Sosman JA, Hodi FS. Survival, durable tumor remission, and long-term safety in patients with advanced melanoma receiving nivolumab. J Clin Oncol. 2014 Apr 1;32(10):1020-30. doi: 10.1200/JCO.2013.53.0105. Epub 2014 Mar 3. PMID 24590637
- [Background] Wang DD, Zhang S, Zhao H, Men AY, Parivar K. Fixed dosing versus body size-based dosing of monoclonal antibodies in adult clinical trials. J Clin Pharmacol. 2009 Sep;49(9):1012-24. doi: 10.1177/0091270009337512. Epub 2009 Jul 20. PMID 19620385
- [Background] Wolchok JD, Kluger H, Callahan MK, Postow MA, Rizvi NA, Lesokhin AM, Segal NH, Ariyan CE, Gordon RA, Reed K, Burke MM, Caldwell A, Kronenberg SA, Agunwamba BU, Zhang X, Lowy I, Inzunza HD, Feely W, Horak CE, Hong Q, Korman AJ, Wigginton JM, Gupta A, Sznol M. Nivolumab plus ipilimumab in advanced melanoma. N Engl J Med. 2013 Jul 11;369(2):122-33. doi: 10.1056/NEJMoa1302369. Epub 2013 Jun 2. PMID 23724867
- [Background] Yuan J, Adamow M, Ginsberg BA, Rasalan TS, Ritter E, Gallardo HF, Xu Y, Pogoriler E, Terzulli SL, Kuk D, Panageas KS, Ritter G, Sznol M, Halaban R, Jungbluth AA, Allison JP, Old LJ, Wolchok JD, Gnjatic S. Integrated NY-ESO-1 antibody and CD8+ T-cell responses correlate with clinical benefit in advanced melanoma patients treated with ipilimumab. Proc Natl Acad Sci U S A. 2011 Oct 4;108(40):16723-8. doi: 10.1073/pnas.1110814108. Epub 2011 Sep 20. PMID 21933959
- [Background] Zhang C, Wu S, Xue X, Li M, Qin X, Li W, Han W, Zhang Y. Anti-tumor immunotherapy by blockade of the PD-1/PD-L1 pathway with recombinant human PD-1-IgV. Cytotherapy. 2008;10(7):711-9. doi: 10.1080/14653240802320237. PMID 18841514
- [Background] Zhang S, Shi R, Li C, Parivar K, Wang DD. Fixed dosing versus body size-based dosing of therapeutic peptides and proteins in adults. J Clin Pharmacol. 2012 Jan;52(1):18-28. doi: 10.1177/0091270010388648. Epub 2011 Jan 13. PMID 21233304
- [Background] Zou W, Chen L. Inhibitory B7-family molecules in the tumour microenvironment. Nat Rev Immunol. 2008 Jun;8(6):467-77. doi: 10.1038/nri2326. PMID 18500231

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Started | 10
Completed | 2
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 9
Age, Continuous [Median (Standard Deviation); unit: years] | 74 (9.33)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 6
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10
ECOG-Performance Status [Median (Full Range); unit: units on a scale] — ECOG Performance Status (0-5) ECOG-PS 0: Fully active, capable of performing all normal activities without restrictions.
  ECOG-PS 1: Restricted in strenuous activity, but able to perform most activities.
  ECOG-PS 2: Restricted in work activities, but can still manage self-care and some activities.
  ECOG-PS 3: Capable of limited self-care, confined to bed more than 50% of the waking hours.
  ECOG-PS 4: Completely disabled and confined to bed, unable to perform self-care.
  ECOG-PS 5: Deceased.
  units on a scale | 2 [1 to 2]

OUTCOME MEASURES:

1. Primary Outcome: Rate of Split Course Chemoradiation Completion
Description: To determine the percentage of poor risk and/or elderly unresectable stage III NSCLC patients who complete split course chemoradiation. Objective will be assessed as a binary endpoint of yes/no completion for each patient.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
Participants | 8

2. Primary Outcome: Number of Cycles of Durvalumab (MEDI4736) Received for Each Treated Patient
Description: To determine the safety and tolerability of durvalumab (MEDI4736) after completion of chemoradiation in this group of patients. Objective will be measured by (a) the number of cycles of durvalumab received for each treated patient and (b) the binary endpoint of discontinuation of durvalumab.
Time Frame: Up to 1 year
Population: These patients all completed split course chemoradiation, and had the opportunity to receive Durvalumab
Measure: Median (Standard Deviation); unit: Cycles
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 8
Cycles | 4 (4.96)

3. Secondary Outcome: One-year Overall Survival (OS)
Description: To determine the 1-year overall survival rate
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
Participants | 8

4. Secondary Outcome: One-year Progression-Free Survival (PFS) According to RECIST 1.1
Description: To determine the 1-year progression-free survival rate based on the EORTC RECIST 1.1 criteria for solid tumors as follows:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
Participants | 5

5. Secondary Outcome: One-Year Loco-regional Progression-free Survival (PFS) According to RECIST 1.1
Description: To determine the 1-year loco-regional progression-free survival rate, based on the EORTC RECIST 1.1 criteria for solid tumors as follows:
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  Partial Response (PR): At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  Progressive Disease (PD): At least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. (Note: the appearance of one or more new lesions is also considered progression).
  Stable Disease (SD): Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
Participants | 5

6. Secondary Outcome: Rate of Grade 3 and 4 Toxicities Assessed by CTCAE v 5.0
Description: To determine rate of grade 3 and 4 toxicities with this regimen in the selected patient population
Time Frame: 1 year
Measure: Number; unit: percentage of patients
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
Number analyzed (Participants) | 10
percentage of patients | 20

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Concurrent, Split Course Chemoradiation Followed by Durvalumab
All-Cause Mortality (participants affected / at risk) | 2/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 5/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Concurrent, Split Course Chemoradiation Followed by Durvalumab (N=10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2023-06-12): https://cdn.clinicaltrials.gov/large-docs/38/NCT04441138/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-19): https://cdn.clinicaltrials.gov/large-docs/38/NCT04441138/SAP_001.pdf
  • Informed Consent Form (2024-01-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04441138/ICF_002.pdf